CLINICAL TRIAL: NCT00497198
Title: An Exploratory Study of MCI-196 for Treatment of Type 2 Diabetes in Randomized, Double-Blind, Parallel-Assignment, Placebo-Controlled Manner
Brief Title: Efficacy and Safety Study of MCI-196 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: General Manager, Clinical Research Department II, Mitsubishi Tanabe Pharma Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCI196-19
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; anion-exchange resin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — cholebine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MCI-196 (Experimental)
  Interventions: Drug: MCI-196
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo of MCI-196 Tablet

INTERVENTIONS:
Drug: MCI-196 — Three tablets of MCI-196 500mg tablet at a time, three times daily, 12 weeks administration (dose in a day: 4500mg)
  Other Names: Colestilan(INN); Colestimide(JAN); CHOLEBINE
  Arms: MCI-196
Drug: Placebo of MCI-196 Tablet — Three tablets of Placebo tablet at a time, three times daily, 12 weeks administration
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy of MCI-196 in patients with Type 2 Diabetes based on the changes in blood glucose-related parameters and safety after 12 weeks administration in double-blind, placebo-controlled manner. And in addition, the changes in lipid-related parameters are examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose fasting blood glucose levels during the observation period are between 130mg/dL and 200mg/dL.
* Patients whose HbA1c is 7.0% or above during the observation period.

Exclusion Criteria:

* Patients with serious cardiac, hepatic or renal complications.
* Patients with serious diabetic complications.
* Patients with complete biliary obstruction or ileus.
* Pregnant, lactating, and probably pregnant patients, and patients who can not agree to contraception.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2005-10; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation

REFERENCES:
- [Result] Kondo K, Kadowaki T. Colestilan monotherapy significantly improves glycaemic control and LDL cholesterol levels in patients with type 2 diabetes: a randomized double-blind placebo-controlled study. Diabetes Obes Metab. 2010 Mar;12(3):246-51. doi: 10.1111/j.1463-1326.2009.01159.x. Epub 2009 Sep 22. PMID 20047620

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Three tablets of Placebo tablet at a time, three times daily, 12 weeks administration
Period: Overall Study
Arm/Group | MCI-196 | Placebo
Started | 92 | 91
Completed | 87 | 86
Not Completed | 5 | 5
Not completed — Adverse Event | 4 | 2
Not completed — Physician Decision | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MCI-196 | Placebo | Total
Number analyzed (Participants) | 92 | 91 | 183
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 55 | 115
  >=65 years | 32 | 36 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 67
  Male | 59 | 57 | 116

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Low Density Lipoprotein Cholesterol(LDL-c) at Week 12
Time Frame: 12 weeks (baseline to week 12)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | MCI-196 | Placebo
Number analyzed (Participants) | 86 | 86
mg/dL | -28.9 (2.0) | -0.2 (2.0)

2. Primary Outcome: Fasting Plasma Glucose at Baseline
Time Frame: 0 weeks
Population: Per protocol set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MCI-196 | Placebo
Number analyzed (Participants) | 86 | 86
mg/dL | 170.2 (21.1) | 168.2 (20.5)

3. Primary Outcome: Change From Baseline in Blood Glucose at Week 12
Time Frame: 12 weeks (baseline to week 12)
Population: Per protocol set; Last observation carried forward
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | MCI-196 | Placebo
Number analyzed (Participants) | 86 | 86
mg/dL | -21.3 (2.2) | 0.8 (2.2)

4. Primary Outcome: Hemoglobin A1c (HbA1c) at Baseline
Time Frame: 0 weeks
Population: Per protocol set
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MCI-196 | Placebo
Number analyzed (Participants) | 86 | 86
percentage | 7.97 (0.72) | 7.94 (0.77)

5. Primary Outcome: Change From Baseline in Hemoglobin A1c(HbA1c) at Week 12
Time Frame: 12 weeks (baseline to week 12)
Population: Per protocol set; Last observation carried forward
Measure: Mean (Standard Error); unit: percentage
Arm/Group | MCI-196 | Placebo
Number analyzed (Participants) | 86 | 86
percentage | -0.70 (0.06) | 0.18 (0.06)

ADVERSE EVENTS:
Time Frame: 1MCI-196: Three tablets of MCI-196 500mg tablet at a time, three times daily, 12 weeks administration (dose in a day: 4500mg) Placebo: Three tablets of Placebo tablet at a time, three times daily, 12 weeks administration
Arm/Group | MCI-196 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/92 | 5/91
Other Adverse Events (participants affected / at risk) | 53/92 | 46/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-196 (N=92) | Placebo (N=91)
Colon polyp (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-196 (N=92) | Placebo (N=91)
Vertigo (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 2
Corneal erosion (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 1 | 0
Episcleritis (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 12 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Faeces hard (Gastrointestinal disorders) | 3 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastritis atrophic (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Acute tonsillitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis Escherichia coli (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 18 | 12
Otitis media (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 1
Tinea pedis (Infections and infestations) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal neoplasma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 1 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 5 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Schamberg's disease (Skin and subcutaneous tissue disorders) | 0 | 1
Arteriosclerosis obliterans (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other